CLINICAL TRIAL: NCT00909779
Title: A Large Simple Safety Study of Arformoterol Tartrate Inhalation Solution in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Safety Study of Arformoterol Tartrate Inhalation Solution in Chronic Obstructive Pulmonary Disease (COPD) Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 091-080
Record Dates: First submitted 2009-05-26; First posted 2009-05-28 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease (COPD); respiratory; long-acting beta agonist (LABA)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arformoterol 15 mcg twice daily (Experimental): Arformoterol 15 mcg twice daily by nebulization. All subjects will be dispensed albuterol HFA metered-dose inhaler (MDI) to be used as needed as rescue medication for bronchospasm and acute treatment of COPD symptoms.
  Interventions: Drug: Arformoterol
- Placebo twice daily (Placebo Comparator): Placebo twice daily by nebulization. All subjects will be dispensed albuterol HFA metered-dose inhaler (MDI) to be used as needed as rescue medication for bronchospasm and acute treatment of COPD symptoms.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arformoterol — Arformoterol Tartrate Inhalation Solution 15 mcg twice daily (BID) for a duration of one year
  Other Names: Brovana
  Arms: Arformoterol 15 mcg twice daily
Drug: Placebo — Placebo inhalation solution, twice daily (BID) for a duration of one year.
  Arms: Placebo twice daily

SUMMARY:
This is a multi-center study to evaluate the long-term safety of arformoterol 15 mcg twice daily (BID) in the treatment of subjects with moderate-to-severe COPD. Study participation will consist of a total of 6 visits over approximately 1 year.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized, placebo-controlled, parallel-group, outpatient, safety study to evaluate the long-term safety of arformoterol 15 mcg twice daily (BID) in the treatment of subjects with moderate-to-severe COPD. The administration of arformoterol in subjects with moderate to severe COPD will not result in a meaningfully greater incidence of respiratory death and COPD exacerbation -related hospitalizations compared to placebo (nebulized saline and non-long-acting beta2-agonist [LABA] COPD standard of care treatments). This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject must give written informed consent, including privacy authorization as well as adherence to concomitant medication withholding periods, prior to participation.
* Females considered not of childbearing potential must be surgically sterile (total hysterectomy, bilateral salpingo oophorectomy, or tubal ligation) or post-menopausal, which is defined as a complete cessation of menstruation for at least 1 year.
* Male and female subjects must be at least 40 years old at the time of consent.
* Subjects must have a pre-established, documented primary clinical diagnosis of non-asthmatic COPD or are referred for diagnosis of non-asthmatic COPD.
* Subjects must have a baseline FEV1 of ≤50% predicted volume at Visits 1 and 2 (pre-dose).
* Subjects must have a FEV1 >0.50 L at either Visit 1 or 2 (pre-dose).
* Subject's respiratory status must be clinically stable.
* Subjects must have a FEV1/forced vital capacity (FVC) ratio of ≤70% at either Visit 1 or 2 (pre-dose).
* Subjects must have had at least 1 COPD exacerbation within the last year (defined as initiation or an increase in the dose of oral steroids or antibiotics for the treatment of COPD).
* Subjects must have a ≥15 pack-year smoking history and a baseline breathlessness severity grade of ≥2 (Modified Medical Research Council [MMRC] Dyspnea Scale Score) at Visit 2.
* Female subjects ≤65 years of age must have a negative serum pregnancy test conducted at Visit 1 prior to randomization. Females of childbearing potential must be using an acceptable method of birth control.
* Subjects' overall health must be sufficiently stable to complete the study requirements based on the screening physical examination (defined as the absence of any clinically relevant abnormalities), medical history, 12-lead ECG, and clinical laboratory values (hematology, serum chemistry and urinalysis), and vital signs (heart rate, respiratory rate, and blood pressure) that have been conducted within 30 days of Visit 2 (randomization). If any of the hematology, chemistry, or urinalysis results are not within the laboratory's reference range, then the subject can be included only if the investigator judges the deviations to be not clinically significant.
* Subjects must have a minimum blood pressure of 105/60 mmHg and a minimum resting pulse of 50 bpm at Screening Visit 1. Subjects who do not meet these criteria at Screening Visit 1 must meet the criteria on the first day of dosing (Day 1) in order to be eligible for the study. Subjects with a medical condition which causes low blood pressure or low heart rate, but, in the opinion of the Principal Investigator or designee the medical condition could resolve, may be rescreened when the condition is resolved.
* Subjects must be willing and able to complete all study questionnaires and logs reliably.
* Subjects must be willing and able to comply with study procedures and visit schedule.
* Subjects must have sufficient understanding of English to complete all questionnaires and logs.

Exclusion Criteria:

* Female subjects who are pregnant or lactating.
* Subjects with a history of asthma, with the exception of asthma diagnosed in childhood.
* Subjects with a blood eosinophil count >5% of total white blood cell count.
* Subjects with a febrile illness within 3 days before Screening.
* Subjects with a malignant neoplasm other than non melanomatous basal cell skin cancer. Subjects with a history of malignancy who have been cancer free for 5 years or more may be enrolled.
* Subjects who are currently using disallowed medications or will be unable to complete the medication washout periods. Subjects taking a prohibited concurrent medication which requires a washout of >30 days may be rescreened when the washout of the prohibited concurrent medication has been met.
* Subjects with life threatening/unstable respiratory status, including upper or lower respiratory tract infection, within the previous 30 days prior to screening.
* Subjects who have had a change in dose or type of any medications for COPD within 2 weeks prior to the screening visit. Subjects not on a stable dose of COPD medications may be rescreened after being on a stable dose for at least 14 days
* Subjects with a chest x ray taken ≤3 months prior to screening that suggests a diagnosis other than COPD (eg, diagnostic of pneumonia, other infection, atelectasis, or pneumothorax or other active/ongoing pulmonary conditions). If there is no chest x ray taken ≤3 months prior to screening, or if recent results are unavailable for review, a chest x ray must be performed prior to visit 2. Subjects with a medical condition that caused the abnormal finding, but, in the opinion of the Principal Investigator or designee the medical condition could resolve, may be rescreened when the condition is resolved
* Subjects with a positive urine drug test during screening.
* Subjects with a known history of alcohol abuse may be enrolled in the study if the subject's current alcohol use does not exceed more than 3 alcoholic beverages per day.
* Subjects whose schedule or travel prevents the completion of all required visits.
* Subjects who are scheduled for inpatient hospitalization or elective surgery (inpatient or outpatient) during the trial. Subjects may be rescreened when the condition is resolved.
* Subjects have participated in an investigational drug study and/or any COPD interventional trial within 30 days prior to screening or who are currently participating in another investigational drug study or COPD interventional trial.
* Subjects with a history of allergic reaction to the study medication or any components of the study medications.
* Subjects who are study site staff members or relatives of study site staff members directly involved in this study.
* Subjects with clinically significant cardiac, (Functional Class III and IV; Objective Class C and D by New York Heart Association [NYHA] Functional Classification),hepatic, renal, gastrointestinal, endocrine, metabolic, neurologic, or psychiatric disorder that may interfere with successful completion of this protocol.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 841 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- United States (73):
  - Jefferson Clinic, Birmingham, Alabama
  - Alabama Clinical Therapeutic, LLC, Birmingham, Alabama
  - Achieve Clinical Research, Brimingham, Alabama
  - Jasper Summit Research, LLC, Jasper, Alabama
  - Chest Critical Care Consultants, Anaheim, California
  - California Research Medical Group, Fullerton, California
  - Integrated Research Group, Riverside, California
  - Quality Control Research Inc., Roseville, California
  - Sockolov and Sockolov APC, Sacramento, California
  - Centers for Clinical Trials of Sacremento, Sacremento, California
  - Institute of HealthCare Assessment, Inc., San Diego, California
  - National Jewish Health, Denver, Colorado
  - Southeast Clinical Research, Chiefland, Florida
  - Tampa Bay Medical Research Inc., Clearwater, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Avail Clinical Research, DeLand, Florida
  - The Lung Clinic, P.A., Kissimmee, Florida
  - DCT, Orlando, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Canton, Georgia
  - Southeast Regional Research Group, Columbus, Georgia
  - Atlanta Pharmaceutical Research, Decatur, Georgia
  - Wellstar Marietta Pulmonary Medicine, Marietta, Georgia
  - Southeast Regional Research Group, Rincon, Georgia
  - Medisphere Medical Research Center, Evansville, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kentucky Lung Clinic, Hazard, Kentucky
  - Bendel Medical Research Center, LLC, Lafayette, Louisiana
  - ClinSite LLC, Ann Arbor, Michigan
  - Clinical Research Institute Inc., Minneapolis, Minnesota
  - Midwest Chest Consultants, Saint Charles, Missouri
  - C.A.R.E. Clinical Research, St Louis, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Delaware Valley Clinical Research, Cherry Hill, New Jersey
  - New York Pulmonary and Clinical Care Associates, PC, New York, New York
  - ENT & Allergy Associates, Newburgh, New York
  - Rochester Clinical Research, Rochester, New York
  - AAIR Research Center, Rochester, New York
  - American Health Research Inc., Charlotte, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - DayStar Clinical Research, Inc., Akron, Ohio
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Arcuri Clinical Research, LLC, Philadelphia, Pennsylvania
  - Biomedical Research Alliance at Hypertension and Nephrology, Pawtucket, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Lowcountry Lung & Critical Care, PA, Charleston, South Carolina
  - Neem Research Group, Inc., Columbia, South Carolina
  - Gaffney Pharmaceutical Research, Gaffney, South Carolina
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - S. Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - CU Pharmaceutical Research, Union, South Carolina
  - Allergy Associates, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - DCT, Arlington, Texas
  - Baylor College of Medicine, Clinical Studies Unit, Ben Taub General Hospital, Houston, Texas
  - VAMC, Houston, Texas
  - Kingwood Research Institute, LLC, Kingwood, Texas
  - Physician PrimeCare Research, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - DCT, Sugar Land, Texas
  - SouthEast Research Institute, Webster, Texas
  - National Clinical Resources, Inc., Provo, Utah
  - Utah Clinical Trials LLC, Salt Lake City, Utah
  - Charlottesville Medical Research Inc., Charlottesville, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Dominion Medical Associates, Richmond, Virginia
  - Pulmonary Associates of Richmond Inc., Richmond, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - Pulmonary Consultants, PLLC, Tacoma, Washington

REFERENCES:
- [Derived] Donohue JF, Ganapathy V, Bollu V, Stensland MD, Nelson LM. Health Status of Patients with Moderate to Severe COPD after Treatment with Nebulized Arformoterol Tartrate or Placebo for 1 Year. Clin Ther. 2017 Jan;39(1):66-74. doi: 10.1016/j.clinthera.2016.11.021. Epub 2016 Dec 20. PMID 28011247
- [Derived] Donohue JF, Hanania NA, Make B, Miles MC, Mahler DA, Curry L, Tosiello R, Wheeler A, Tashkin DP. One-year safety and efficacy study of arformoterol tartrate in patients with moderate to severe COPD. Chest. 2014 Dec;146(6):1531-1542. doi: 10.1378/chest.14-0117. PMID 25451347

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Twice Daily | Arformoterol 15 Mcg Twice Daily
Started | 421 | 420
Completed | 211 (All subjects but 47 were followed for 12 months/until death (whichever was earlier).) | 255 (All subjects but 42 were followed for 12 months/until death (whichever was earlier).)
Not Completed | 210 | 165
Not completed — Adverse Event | 53 | 55
Not completed — Lack of Efficacy | 7 | 4
Not completed — Lost to Follow-up | 19 | 15
Not completed — Physician Decision | 8 | 2
Not completed — Protocol Violation | 2 | 5
Not completed — Withdrawal by Subject | 116 | 80
Not completed — Site Ceasing Operation | 2 | 2
Not completed — Medical Monitor Decision | 1 | 0
Not completed — Noncompliance | 1 | 1
Not completed — Randomized in error | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Comparator: Placebo Twice Daily: Placebo twice daily by nebulization. All subjects will be dispensed albuterol HFA metered-dose inhaler (MDI) to be used as needed as rescue medication for bronchospasm and acute treatment of COPD symptoms.
- Experimental: Arformoterol 15 Mcg Twice Daily: Arformoterol 15 mcg twice daily by nebulization. All subjects will be dispensed albuterol HFA metered-dose inhaler (MDI) to be used as needed as rescue medication for bronchospasm and acute treatment of COPD symptoms.
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator: Placebo Twice Daily | Experimental: Arformoterol 15 Mcg Twice Daily | Total
Number analyzed (Participants) | 421 | 420 | 841
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 222 | 204 | 426
  >=65 years | 199 | 216 | 415
Age Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.5) | 64.2 (9.3) | 63.8 (9.4)
Sex/Gender, Customized [Number; unit: participants]
  Female | 178 | 183 | 361
  Male | 243 | 236 | 479
  Undifferentiated | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 9 | 24
  Not Hispanic or Latino | 402 | 411 | 813
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 45 | 88
  White | 374 | 372 | 746
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 421 | 420 | 841
Number of COPD exacerbations in last year [Mean (Standard Deviation); unit: Number of occurrences] — The average number of COPD exacerbations during the previous year
  Number of occurrences | 0.8 (1.1) | 1.0 (1.4) | 0.9 (1.3)
FEV1 [Mean (Standard Deviation); unit: Liter] — FEV1: Forced expiratory volume in one second. FEV1 was measured at Visit 1 (screening), pre- and post-albuterol administration for reversibility testing, pre-dose at Visits 2 through 5, and at Visit 6/EOS. The best FEV1 from at least 3 acceptable maneuvers was recorded. Study baseline was defined as the Visit 2 pre-dose value. If the Visit 2 pre-dose value was missing, the last FEV1 value obtained prior to first treatment was used for baseline.
  Liter | 1.178 (0.487) | 1.176 (0.482) | 1.177 (0.485)
Percent predicted FEV1 (%) [Mean (Standard Deviation); unit: Percentage (%)] — Best FEV1 percent predicted was measured at Visit 1 (screening), pre-dose at Visits 2 through 5, and at Visit 6/EOS, as described for FEV1.
  Percentage (%) | 39.4 (13.9) | 39.7 (13.2) | 39.5 (13.5)
Baseline smoking status [Number; unit: Current] — Smoking status was recorded at each visit. At baseline, a subject was only defined as a former smoker if they had given up smoking at least 6 calendar months prior to the Visit 1 (screening) date based on the smoking cessation date. Otherwise, they were classified as a current smoker.
  Current
    Current | 218 | 214 | 432
    Former | 203 | 206 | 409
Number of pack-years smoked [Number; unit: Pack-years] — Number of pack-years smoked was defined as the number of cigarette packs smoked per day times the number of years smoked.
  Pack-years
    ≥ 15 - < 25 | 41 (9.7) | 40 (9.5) | 81 (9.6)
    ≥ 25 - < 30 | 36 (8.6) | 29 (6.9) | 65 (7.7)
    ≥ 30 | 344 (81.7) | 351 (83.6) | 695 (82.6)
Baseline Oral/Inhaled Corticosteroid Use [Number; unit: participants] — Oral or inhaled corticosteroid use
  participants
    No | 202 (48.0) | 202 (48.1) | 404 (48.0)
    Yes | 219 (52.0) | 218 (51.9) | 437 (52.0)
Baseline Oxygen Therapy Use [Number; unit: participants] — Oxygen therapy use at baseline
  participants
    No | 330 (78.4) | 334 (79.5) | 664 (79.0)
    Yes | 91 (21.6) | 86 (20.5) | 177 (21.0)

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Respiratory Death or First COPD Exacerbation Related Hospitalization (Whichever Occurs First).
Description: COPD exacerbation: an increase in COPD symptoms that necessitated any change in baseline medication (bronchodilators,anti-inflammatory agents, antibiotics, supplemental oxygen therapy, etc.).Hospitalization: any inpatient admission or any emergency department visit > 24 hours in duration. Hospice was considered hospitalization.COPD exacerbation related hospitalization: hospitalization that was due to 1) COPD exacerbation or 2) a COPD exacerbation preceded, or occurred concomitantly with the onset of, the event for which the subject was hospitalized.Respiratory-related death: For each death the Primary Investigator designated a 'probable cause', which was the primary condition that precipitated the terminal events that were the immediate cause of death. If a probable cause could not be ascertained, the cause of death was considered 'UNKNOWN'. Cause other than 'UNKNOWN' was categorized as either respiratory or non-respiratory. Deaths of 'UNKNOWN' cause were counted as primary events.
Time Frame: 0-12 months
Population: Intent-to-treat population: subjects who were randomized to treatment and received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Subjects with Primary Event
Groups:
- Placebo: Placebo twice daily
Arm/Group | Experimental: Arformoterol 15 Mcg Twice Daily | Placebo
Number analyzed (Participants) | 420 | 421
Number analyzed (Subjects with Primary Event) | 63 | 40
Days | 155.0 (91.2) [0.425 to 0.864] | 171.7 (98.7)
Statistical Analysis 1: Comparison: Experimental: Arformoterol 15 Mcg Twice Daily; The null hypothesis is: There is 40% or higher excess risk of the primary events in the arformoterol group relative to placebo (a constant hazard ratio of 1.4). The primary analysis was a Cox proportional hazards regression model, with treatment group, baseline smoking status, sex, age, BMI, and baseline FEV1 as covariates. The hazard ratio and 90% two-sided confidence interval for the hazard ratio (adjusted for the interim analysis) comparing arformoterol to placebo were estimated; Test type: Non-Inferiority or Equivalence — The study was powered under a one-sided alternative hypothesis, in which arformoterol is superior to placebo, with a hazard ratio of 0.80 or less. To achieve 80% power, it was necessary to observe 86 total events for the primary endpoint adjusted for interim analysis. Assuming an annual event proportion of 17.3% in the placebo group and 30% lost to follow-up, we anticipated to randomize approximately 900 subjects (450 per arm). The non-inferiority margin for the hazard ratio is 1.4; Regression, Cox; Hazard Ratio (HR) = 0.606, 95% CI 2-sided [0.425 to 0.864] — Hazard ratio was calculated as arformoterol vs. placebo

2. Secondary Outcome: The Incidence of Protocol Defined COPD Exacerbations.
Description: A protocol-defined exacerbation of COPD was defined as an increase in respiratory symptoms (classically, increased shortness of breath, increased sputum production, and/or increased sputum purulence) that necessitates any change in baseline medication other than bronchodilators (e.g., anti-inflammatory agents, antibiotics, supplemental oxygen therapy, etc) or causes the subject to require additional medical attention (i.e., emergency room visit or hospitalization).
Time Frame: 0-12 months
Population: Intent-to-treat population: subjects who were randomized to treatment and received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Placebo Comparator: Placebo Twice Daily: Placebo twice daily by nebulization. All subjects will be dispensed albuterol HFA metered-dose inhaler (MDI) to be used as needed as rescue medication for bronchospasm and acute treatent of COPD symptoms.
Arm/Group | Placebo Comparator: Placebo Twice Daily | Experimental: Arformoterol 15 Mcg Twice Daily
Number analyzed (Participants) | 421 | 420
participants
  Overall | 132 | 122
  1 COPD event | 72 | 71
  2 COPD events | 34 | 29
  3 or more COPD events | 26 | 22

3. Secondary Outcome: The Incidence of All Cause Mortality
Description: Survival status at the end of the study will be determined for each subject. The proportion of subjects dead and the annual event rate will be summarized by treatment.
Time Frame: 0-12 months
Population: Intent-to-treat population: subjects who were randomized to treatment and received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo Comparator: Placebo Twice Daily | Experimental: Arformoterol 15 Mcg Twice Daily
Number analyzed (Participants) | 421 | 420
participants | 10 | 12

4. Secondary Outcome: The Incidence of Treatment Emergent AEs
Description: TEAEs were defined as: 1) adverse events that occurred on or after the date of first dose of study medication, 2) adverse events with a missing start date and a stop date on or after the date of first does of study medication, or 3) adverse events with both a missing start and stop date.
  The frequency and percentage of subjects with TEAEs were summarized. At each level of summarization, a subject was counted only once for each AE he/she experienced within that level. The percentage of subjects having had at least 1 AE at each level was calculated.
Time Frame: 0-12 months
Population: Intent-to-treat population: subjects who were randomized to treatment and received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo Comparator: Placebo Twice Daily | Experimental: Arformoterol 15 Mcg Twice Daily
Number analyzed (Participants) | 421 | 420
participants | 287 | 306

5. Secondary Outcome: SGRQ: Mean Change From Baseline in Total Score
Description: The SGRQ assessed health status and consisted of 3 component scores (Symptoms, Activity, and Impacts) as well as a total score. Items were scored in accordance with the developer's guidelines. Scores were expressed as a percentage of overall impairment, where 100 represented worst possible health status and 0 indicated best possible health status. The SGRQ was assessed pre-dose at baseline, months 3, 6 and 12 or the end of study (EOS). Visit 2 was defined as baseline. A change from baseline in the Total Score of ≥ 4 units is considered the minimal clinically important difference (MCID) for SGRQ.
Time Frame: Baseline and on treatment at months 3, 6 and 12 (or early termination)
Population: Intent-to-treat population: subjects who were randomized to treatment and received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Placebo Comparator: Placebo Twice Daily | Experimental: Arformoterol 15 Mcg Twice Daily
Number analyzed (Participants) | 421 | 420
Score
  Month 3 (n=276,308) | -1.544 (0.609) | -3.876 (0.575)
  Month 6 (n=233,287) | -1.855 (0.746) | -4.054 (0.679)
  Month 12 (n=199,236) | -2.673 (0.800) | -4.796 (0.735)
  EOS (n=375,379) | -0.587 (0.616) | -3.231 (0.613)

6. Secondary Outcome: FEV1: Mean Change From Baseline
Description: FEV1 was measured at Visit 1 (screening), pre- and post-albuterol administration for reversibility testing, pre-dose at baseline, months 3, 6, 9 and 12/EOS. The best FEV1 from at least 3 acceptable maneuvers was recorded. Study baseline was defined as the Visit 2 pre-dose value. If the Visit 2 pre-dose value was missing, the last FEV1 value obtained prior to first treatment was used for baseline.
Time Frame: Baseline and on treatments at months 3, 6, 9 and 12 (or early termination)
Population: Intent-to-treat population: subjects who were randomized to treatment and received at least 1 dose of study medication.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo Comparator: Placebo Twice Daily | Experimental: Arformoterol 15 Mcg Twice Daily
Number analyzed (Participants) | 421 | 420
Liter
  Month 3 (n=289,331) | 0.027 (0.018) | 0.093 (0.016)
  Month 6 (n=248,300) | 0.036 (0.023) | 0.090 (0.021)
  Month 9 (n=223,268) | 0.048 (0.019) | 0.092 (0.018)
  Month 12 (n=206,253) | 0.020 (0.020) | 0.059 (0.018)
  EOS (n=380,391) | 0.047 (0.016) | 0.072 (0.016)

7. Secondary Outcome: Percent Predicted FEV1: Mean Change From Baseline
Description: Percent predicted FEV1: measured FEV1 as a percent of the "predicted values" for the patients of similar characteristics (height, age, sex, and sometimes race and weight). Best FEV1 percent predicted was measured at Visit 1 (screening), pre-dose at baseline, months 3, 6, 9 and 12/EOS, as described for FEV1.
Time Frame: Baseline and on treatments at months 3, 6, 9 and 12 (or early termination)
Population: Intent-to-treat population: subjects who were randomized to treatment and received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo Comparator: Placebo Twice Daily | Experimental: Arformoterol 15 Mcg Twice Daily
Number analyzed (Participants) | 421 | 420
Liter
  Month 3 (n=289,331) | 1.410 (0.533) | 3.480 (0.498)
  Month 6 (n=248,300) | 1.768 (0.648) | 3.460 (0.594)
  Month 9 (n=223,268) | 2.606 (0.626) | 3.651 (0.576)
  Month 12 (n=206,252) | 1.678 (0.642) | 2.662 (0.586)
  EOS (n=380,391) | 2.156 (0.493) | 2.936 (0.486)

8. Secondary Outcome: Forced Vital Capacity (FVC): Mean Change From Baseline
Description: Forced Vital capacity: the volume of air that can forcibly be blown out after full inspiration. Best FVC was measured at Visit 1 (screening), pre-dose at baseline, months 3, 6, 9 and 12/EOS. The best FVC from at least 3 acceptable maneuvers was recorded.
Time Frame: Baseline and on treatment at months 3, 6, 9 and 12 (or early termination)
Population: Intent-to-treat population: subjects who were randomized to treatment and received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo Comparator: Placebo Twice Daily | Experimental: Arformoterol 15 Mcg Twice Daily
Number analyzed (Participants) | 421 | 420
Liter
  Month 3 (n=289,331) | 0.039 (0.024) | 0.139 (0.022)
  Month 6 (n=248,300) | 0.056 (0.031) | 0.120 (0.028)
  Month 9 (n=223,268) | 0.049 (0.029) | 0.139 (0.027)
  Month 12 (n=206,253) | 0.040 (0.029) | 0.088 (0.027)
  EOS (n=380,391) | 0.056 (0.022) | 0.102 (0.022)

9. Secondary Outcome: Inspiratory Capacity (IC): Mean Change From Baseline
Description: IC: the total amount of air that can be drawn into the lungs after normal expiration.
  IC was measured pre- and post-albuterol administration at Visit 1 (screening), pre-dose at baseline, months 3, 6, 9 and 12/EOS. IC maneuvers were done in triplicate. The mean of all recorded IC values was used for each subject at each time point. Study baseline was defined as the Visit 2 pre-dose value. If the Visit 2 pre-dose value was missing, the last IC value obtained prior to first treatment dose was used for baseline.
Time Frame: Baseline and on treatment at months 3, 6, 9 and 12 (or early termination)
Population: Intent-to-treat population: subjects who were randomized to treatment and received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo Comparator: Placebo Twice Daily | Experimental: Arformoterol 15 Mcg Twice Daily
Number analyzed (Participants) | 421 | 420
Liter
  Month 3 (n=284,320) | 0.030 (0.023) | 0.054 (0.021)
  Month 6 (n=243,298) | -0.011 (0.026) | 0.067 (0.024)
  Month 9 (n=218,258) | 0.046 (0.029) | 0.096 (0.027)
  Month 12 (n=199,246) | 0.004 (0.029) | 0.035 (0.027)
  EOS (n=374,384) | 0.031 (0.022) | 0.058 (0.021)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Placebo Comparator: Placebo Twice Daily | Experimental: Arformoterol 15 Mcg Twice Daily
Serious Adverse Events (participants affected / at risk) | 95/421 | 86/420
Other Adverse Events (participants affected / at risk) | 180/421 | 174/420
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator: Placebo Twice Daily (N=421) | Experimental: Arformoterol 15 Mcg Twice Daily (N=420)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 3 (3)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Corpulmonale (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 3 (3)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (2)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 9 (10) | 3 (4)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastritis fungal (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis bacteria (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomy (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1)
Peridiverticular abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 14 (18) | 12 (13)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 1 (4) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 55 (76) | 35 (44)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator: Placebo Twice Daily (N=421) | Experimental: Arformoterol 15 Mcg Twice Daily (N=420)
Bronchitis (Infections and infestations) | 28 (36) | 43 (58)
Nasopharyngitis (Infections and infestations) | 33 (49) | 38 (50)
Sinusitis (Infections and infestations) | 22 (29) | 19 (27)
Upper respiratory tract infection (Infections and infestations) | 22 (26) | 22 (28)
Headache (Nervous system disorders) | 21 (39) | 35 (53)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 83 (122) | 75 (115)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (46) | 24 (27)

LIMITATIONS AND CAVEATS:
Although LABAs other than study medication were discontinued, other medications were not controlled for. A large number of subjects discontinued after a primary event and their eventual outcomes are unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.